CLINICAL TRIAL: NCT03518541
Title: Controlling Femoral Derotation Osteotomy In Cerebral Palsy With Electromagnetic Tracking - A Randomized Controlled Trial
Brief Title: Controlling Femoral Derotation Osteotomy In Cerebral Palsy With Electromagnetic Tracking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Else Kröner Fresenius Foundation (Other)
Responsible Party: Principal Investigator, Thomas Dreher, Prof. Dr. med. Thomas Dreher, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: InstruFDO
Record Dates: First submitted 2017-12-20; First posted 2018-05-08 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Gait Disorders, Neurologic; Cerebral Palsy; Malalignment
MeSH Terms: conditions — Gait Disorders, Neurologic; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomization into two study arms:
  1. Classic control of derotation using a Moeltgen goniometer intraoperatively
  2. Control of derotation using an electromagnetic tracking device intraoperatively
Who Masked: Participant
Masking Description: Patients are masked about which group they are randomized in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goniometer (Active Comparator): FDO: classic procedure with goniometer controlled derotation
  Interventions: Procedure: Femoral Derotation Osteotomy (FDO)
- EMT (Experimental): FDO: procedure with electromagnetic tracking (EMT) controlling derotation
  Interventions: Procedure: Femoral Derotation Osteotomy (FDO)

INTERVENTIONS:
Procedure: Femoral Derotation Osteotomy (FDO) — Correction of malrotation of the femoral bone by osteotomy, derotation and osteosynthesis

SUMMARY:
The study is designed to evaluate the use of electromagnetic tracking in transversal plane femoral derotation osteotomies. The goal is to raise the precision of the surgical procedure in order to improve the outcome in short- and long term. All patients are examined with an instrumented 3D gait analysis pre- and one year postoperatively. The electromagnetic tracking system is evaluated against a base line CT or MRI scan serving as reference standard pre- and postoperatively.

DETAILED DESCRIPTION:
Internal rotation gait is a common deformity in children, especially in those with spastic diplegia. The treatment includes soft tissue and bony correction. Especially the bony procedures e.g. femoral derotation osteotomies have proven to be effective both in short term and long term evaluation. Nonetheless there is still a relevant number of patients that suffer from over- or under-correction and recurrence over time. The reasons are diverse and include false measurement of the derotation in OR.

The study now evaluates electromagnetic tracking for femoral derotation to improve these results.

The patients are recruited from the outpatients department and included if they meet the criteria.

A baseline rotational CT or MRI scan and a 3D gait analysis are performed preoperatively. The patients are randomized into a electromagnetic tracking group or a classical goniometer group. The derotation is measured with the EMT system or with a classic Moeltgen goniometer in the OR. Goal is to achieve the planned amount of derotation more accurately.

The surgical procedure follows standard rules and does not need alterations because of the study.

After the operation a second rotational CT or MRI scan is performed and the derotation precisely evaluated by two raters and later compared to the results of the intraoperative electromagnetic tracking system. One year postoperative a second 3D gait analysis is performed to measure and compare the functional and dynamic outcome.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy
* GMFCS level I-III
* Functionally disturbing internal rotation gait
* Indication for femoral derotation osteotomy

Exclusion Criteria:

* No capacity of consent
* Inability to perform all needed types examinations
* Minors: Inability of getting a MRI rotational scan (i.e. pacemaker)

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparing the mean hip rotation between the groups | One year after surgery
  Measuring the functional outcome with the mean hip rotation in stance comparing pre- and postoperative gait analysis .
Comparing the mean pelvic rotation between the groups | One year after surgery
  Measuring the functional outcome with the mean pelvic rotation comparing pre- and postoperative gait analysis .

SECONDARY OUTCOMES:
Evaluate actual amount of bony derotation | Shortly after surgery (not ore than 3 month) and again one year after surgery
  Measuring the actual amount of derotation in degrees in a postoperative CT or MRI scan, given in degrees.
Comparing the bony derotation between the groups | Shortly after surgery (not ore than 3 month) and again one year after surgery
  Comparing the planned amount of derotation in degrees with the intraoperative electromagnetic tracking values and the postoperative rotational MRI values in degrees to evaluate the accuracy of implementing a certain amount of bony derotation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dreher, Prof. Dr., Study Director — University Hospital Heidelberg
Locations (1):
- Orthopedic Department, University of Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Geisbusch A, Auer C, Dickhaus H, Putz C, Dreher T. Electromagnetic tracking for femoral derotation osteotomy-an in vivo study. J Orthop Res. 2017 Dec;35(12):2652-2657. doi: 10.1002/jor.23579. Epub 2017 May 23. PMID 28419537
- [Background] Geisbusch A, Auer C, Dickhaus H, Niklasch M, Dreher T. Electromagnetic bone segment tracking to control femoral derotation osteotomy-A saw bone study. J Orthop Res. 2017 May;35(5):1106-1112. doi: 10.1002/jor.23348. Epub 2016 Jul 4. PMID 27325569